CLINICAL TRIAL: NCT00624624
Title: Follow-up of Serum Androgen Profile After Bariatric Surgery in Men With Obesity Related Hypogonadotropic Hypogonadism
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Other Study IDs: LTC-472-120607
Record Dates: First submitted 2008-02-15; First posted 2008-02-27 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Morbid Obesity; Hypogonadism
Keywords: hypogonadotropic hypogonadism; bariatric surgery; serum androgen levels; bone density
MeSH Terms: conditions — Obesity, Morbid; Hypogonadism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Eugonadal men with "Lapband"
- 2: Hypogonadal men with "Lapband"
- 3: Eugonadal men with gastric bypass procedure
- 4: Hypogonadal men with gastric bypass procedure

SUMMARY:
The purpose of this study is to determine the natural course of the androgen profile after bariatric surgery in men with obesity related hypogonadotropic hypogonadism.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 20-55 years
* Planned bariatric procedure
* Helicobacter pylori negative or adequate HP eradication

Exclusion Criteria:

* Liver and/or kidney dysfunction
* Psychiatric disease
* Medication influencing androgen profile and/or bone metabolism
* Weight > 160 kg

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Men with planned bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H de Boer, MD, PhD, Principal Investigator — Rijnstate Hospital
Locations (1):
- Rijnstate Hospital, Arnhem, Netherlands